CLINICAL TRIAL: NCT05705778
Title: Prognostic Value of Plasma Biomarkers Among Patients With Amblyopia
Brief Title: Plasma Biomarker in Amblyopia Patients
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Jingrong Li, Professor, Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2022KYPJ102
Record Dates: First submitted 2022-12-19; First posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Amblyopia
Keywords: amblyopia; plasma biomarker; prediction; treatment outcome
MeSH Terms: conditions — Amblyopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Strabismic
  Interventions: Procedure: standard amblyopia treatment
- Anisometropic
  Interventions: Procedure: standard amblyopia treatment
- Isoametropic
  Interventions: Procedure: standard amblyopia treatment
- Visual deprivation
  Interventions: Procedure: standard amblyopia treatment
- Mixed group
  Interventions: Procedure: standard amblyopia treatment

INTERVENTIONS:
Procedure: standard amblyopia treatment — amblyopia treatment following international guidelines and genetic tests.
  Other Names: plasma biomarker test

SUMMARY:
This prospective study aims to observe the predictive effect of peripheral blood plasma biomarker on the outcome of treatment in children with different types of amblyopia. We also investigated the mechanism of neuromodulation in the visual development of amblyopic children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with amblyopia
* 3-12 years of age
* Able to tolerate amblyopia treatment
* Agree to be involved in this study and agree to have a follow up visit every 3 months.

Exclusion Criteria:

* Have previous treatment history before
* Have pathological ocular anomalies known to cause reduced visual acuity
* Have previous psychiatric, visual or neurological disorders
* Have eccentric fixation and/or abnormal retinal correspondence
* Have attention disorder and learning disability that cannot comprehend psychophysical test instructions given and/or consent for themselves

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: amblyopia patients
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Plasma protein predictor screening for visual acuity improvement following amblyopia therapy using Tandem Mass Tags proteomics | 2 years after including into this clinical trial
  Peripheral blood will be collected prior and after treatment. The plasma will be separated and Tandem Mass Tags will be used for proteomics. We will detect the different expression of plasma protein between successfully treated and untreated amblyopia patients to find biomarkers that predict amblyopia treatment success. Amblyopia treatment success is defined as best corrected visual acuity (BCVA) improvement of 3 or more logMAR lines.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No